CLINICAL TRIAL: NCT02693769
Title: A Randomised, Single Blind, Cross-over Study to Compare a Fixed Dose Combination of Fluticasone Propionate / Formoterol Fumarate (Breath Actuated Inhaler (BAI)) With a Fixed Dose Combination of Indacaterol Maleate / Glycopyrronium Bromide (Ultibro® Breezhaler) in Subjects With Fixed Airflow Obstruction and Elevated Eosinophils
Brief Title: A Study to Compare Fluticasone /Formoterol Breath Actuated Inhaler (BAI) and Ultibro in Subjects With Fixed Airflow Obstruction and Elevated Eosinophils
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KFL3503
Record Dates: First submitted 2016-02-08; First posted 2016-02-29 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-08

CONDITIONS: ACOS (Fixed Airflow Obstruction and Elevated Eosinophils)
MeSH Terms: interventions — Fluticasone; Glycopyrrolate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone/formoterol BAI (Experimental): To compare the efficacy of fluticasone/formoterol BAI 125/5 μg (2 puffs b.i.d.)
  Interventions: Drug: fluticasone propionate/formoterol fumarate breath actuated inhaler; Drug: Indacaterol maleate / glycopyrronium bromide capsules
- Ultibro Breezhaler (Active Comparator): Ultibro Breezhaler 85/43 µg (1 puff o.d.)
  Interventions: Drug: fluticasone propionate/formoterol fumarate breath actuated inhaler; Drug: Indacaterol maleate / glycopyrronium bromide capsules

INTERVENTIONS:
Drug: fluticasone propionate/formoterol fumarate breath actuated inhaler
Drug: Indacaterol maleate / glycopyrronium bromide capsules

SUMMARY:
The purpose of this study is to investigate whether fluticasone/formoterol Breath actuated inhaler is effective and well tolerated in the treatment of subjects with fixed airflow obstruction and elevated eosinophils.

DETAILED DESCRIPTION:
The study is designed to provide efficacy and safety data for the use of fluticasone/formoterol Breath actuated inhaler in subjects with the characteristics of fixed airflow obstruction and elevated eosinophils. These patients have typically been excluded from previous Flutiform pMDI asthma and chronic obstructive pulmonary disease (COPD) trials; for example in asthma studies, patients with a smoking history of 10 pack years or more have been excluded, conversely in COPD studies patients with any prior history of asthma have been excluded. It is expected that the data from this study will provide a greater understanding of the effects of fluticasone/formoterol in this patient population

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 40 years at Screening visit.
2. Adequate contraception:
3. Diagnosis of fixed airflow obstruction with elevated eosinophils
4. Subjects symptomatic at Visit 1 (CAT ≥10) despite currently receiving treatment with either LAMA or LABA monotherapy or LAMA + LABA as a combination inhaler or separate inhalers.
5. Documented history of ≥ 1 moderate or severe respiratory disease exacerbations (requiring treatment with systemic corticosteroids and/or antibiotics and/or hospitalisation) in the previous year.
6. Willing and able to replace current therapy for obstructive lung disease with study medication.
7. Able to demonstrate correct use of a BAI, Breezehaler and pMDI.

Exclusion Criteria:

1. Respiratory disease exacerbation between 4 weeks prior to screening and Visit 3 (Randomisation).
2. Previous treatment with ICS.
3. Documented evidence of α1-antitrypsin deficiency.
4. Other active respiratory disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung disease, cystic fibrosis, bronchiolitis obliterans.
5. Use of long-term oxygen therapy (LTOT) at least 12 hours daily or mechanical ventilation.
6. Chest X-ray or CT scans performed prior to screening which reveal evidence of clinically significant abnormalities reflective of active disease not believed to be due to COPD
7. Evidence of uncontrolled cardiovascular disease.
8. Evidence of clinically significant renal, hepatic, gastrointestinal, or psychiatric disease.
9. Current malignancy or a previous history of cancer which has been in remission for < 5 years (basal cell or squamous cell carcinoma of the skin which has been resected is not excluded).
10. Clinically significant sleep apnoea requiring use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device.
11. Participation in the acute phase of a pulmonary rehabilitation programme within 4 weeks prior to screening or during the study.
12. Known or suspected history of drug or alcohol abuse in the last 2 years.
13. Requiring treatment with any of the prohibited concomitant medications.
14. Known or suspected hypersensitivity or contraindication to any of the study drugs or excipients.
15. Received an investigational drug within 30 days of the Screening.
16. Received a systemic corticosteroid within 30 days of the Screening visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of fluticasone/formoterol BAI 125/5 μg (2 puffs b.i.d.) versus Ultibro Breezhaler 85/43 µg (1 puff o.d.) in terms of the percentage of eosinophils in induced sputum | at Week 6 of each treatment

SECONDARY OUTCOMES:
The efficacy of fluticasone/formoterol BAI 125/5 μg (2 puffs b.i.d.) versus Ultibro Breezhaler 85/43 µg (1 puff o.d.) in terms of the serum concentration of surfactant protein D (SPD) | at Week 6 of each treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- JURMED, s.r.o., Košice, Slovakia